CLINICAL TRIAL: NCT01098136
Title: A Study of Pelvic Girdle Pain in a Pregnant Population in Western Norway - Incidence, Cumulative Prevalence, Course and Intervention.
Brief Title: Pelvic Girdle Pain in a Pregnant Population in Western Norway.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University of Stavanger (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/174-4
Record Dates: First submitted 2010-03-22; First posted 2010-04-02 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Pelvic Girdle Pain
Keywords: Pelvic girdle pain; Chiropractic; Single-blinded; Outcome study
MeSH Terms: conditions — Pelvic Girdle Pain | interventions — Manipulation, Chiropractic; Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chiropractic treatment (Active Comparator): Management for one-sided pelvic pain, as decided by the chiropractor
  Interventions: Other: Chiropractic
- Conventional health care (Active Comparator): Conventional health care for one-sided pelvic pain
  Interventions: Other: Conventional medical intervention
- Conventional and alternative treatment (Active Comparator): Treament of pregnant women with other pelvic pain syndromes.
  Interventions: Other: Conventional and alternative intervention

INTERVENTIONS:
Other: Chiropractic — Manual treatment of musculoskeletal complaints
  Arms: Chiropractic treatment
Other: Conventional medical intervention — Medical, physiotherapy
  Arms: Conventional health care
Other: Conventional and alternative intervention — Medical and alternative methods for treatment of pelvic pain syndromes
  Arms: Conventional and alternative treatment

SUMMARY:
The objectives in this study are

1. to explore the incidence and cumulative prevalence of pelvic girdle pain (PGP) and its subgroups in a prospective longitudinal study during pregnancy, from 18 weeks until 6 weeks after delivery.
2. to examine the outcome of chiropractic management for a dominating one-sided PGP subgroup of pregnant women in a single-blinded controlled study, and to use efficacy measures that include pain, functional impairment, and sick-leave frequency.
3. to investigate possible predictors for treatment outcome in one-sided PGP in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Lumbopelvic pain
* Pelvic pain
* Performed ultrasound examination at 18th pregnancy week
* Expected normal pregnancy without complications
* Good competency in Norwegian language

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
P4/thigh thrust | Outcome is assessed at follow-up examination 6 weeks post-partum
  As outcome measures we are using pain provocation tests (P4/thigh thrust, Patrick's Faber, Gaenslen's test, and modified Trendelenburg's test), pain palpation tests (long dorsal ligament test and palpation of the symphysis), and a functional test, the active straight leg raise (ASLR) test. All tests are published and described in European guidelines on pelvic girdle pain (PGP). Vleeming A, Albert HB, Ostgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. Eur Spine J. 2008 Jun;17(6):794-819. Epub 2008 Feb 8.

SECONDARY OUTCOMES:
Oswestry Disability Index | Outcome is assessed at follow-up examination 6 weeks post-partum
  The Oswestry Disability Index is one of the principal condition-specific outcome measures the last 30 years for management of disabling effects from spinal disorders

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Malmquist, DC MSc, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Department of Obstetrics and Gynaecology, Stavanger, Norway

REFERENCES:
- [Derived] Gausel AM, Kjaermann I, Malmqvist S, Andersen K, Dalen I, Larsen JP, Okland I. Chiropractic management of dominating one-sided pelvic girdle pain in pregnant women; a randomized controlled trial. BMC Pregnancy Childbirth. 2017 Sep 29;17(1):331. doi: 10.1186/s12884-017-1528-9. PMID 28962596